CLINICAL TRIAL: NCT01249196
Title: A Confirmatory Trial of SK-PC-B70M in Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMART_AD_III_2009
Record Dates: First submitted 2010-11-23; First posted 2010-11-29 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2010-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SK-PC-B70M

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: SK-PC-B70M
- SK-PC-B70M 200mg bid (Experimental)
  Interventions: Drug: SK-PC-B70M
- SK-PC-B70M 300mg bid (Experimental)
  Interventions: Drug: SK-PC-B70M
- Donepezil (Other)
  Interventions: Drug: SK-PC-B70M

INTERVENTIONS:
Drug: SK-PC-B70M — for dosage

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SK-PC-B70M in patients with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable Alzheimer's disease(DSM-IV and NINCDS-ADRDA criteria)
* MRI within the last 12 months consistent with a diagnosis of AD
* MMSE score of 10 to 26 and CDR of 1 or 2
* AChEI or memantine was not taken at least 3 months prior to screening

Exclusion Criteria:

* Other central nervous disease
* Hypothyroidism, Vitamin B12/ Folic acid deficiency, Hypercalcemia, Neurosyphilis, AIDS
* T.I.A or Major infarction within the last 12 months
* Any serious disorder that could limit the ability of the patient to participate in the study
* COPD or asthma
* Any condition which would make the patient or the caregiver, in the opinion of the investigator, unsuitable for the study

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
ADAS-cog (Alzheimer's Disease Assessment Scale-cognitive subscale) | 30 minutes

SECONDARY OUTCOMES:
CIBIC-Plus (Clinician's Interview-Based Impression of Change-Plus caregiver input) | 45 minutes
MMSE (Mini Mental State Examination) | 10 minutes
CDR-SB (Clinical Dementia Rating Sum of Box) | 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- SKChemicals invetigational site, Seoul, South Korea